CLINICAL TRIAL: NCT03090126
Title: Assessment of Therapeutic Education About Non Invasive Ventilation in Patients With Chronic Respiratory
Brief Title: Assessment of Therapeutic Education About Non Invasive Ventilation in Patients With Chronic Respiratory Failure (QoVNI)
Acronym: QoVNI
Status: Withdrawn | Type: Observational
Why Stopped: No possibility to recruit.
Sponsor: Association pour le Développement et l'Organisation de la Recherche en Pneumologie et sur le Sommeil (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-A00189-44
Record Dates: First submitted 2017-03-15; First posted 2017-03-24 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Alveolar Hypoventilation
MeSH Terms: conditions — Hypoventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Alveolar hypoventilation
  Interventions: Other: Therapeutic education

INTERVENTIONS:
Other: Therapeutic education — Questionnaires

SUMMARY:
The purpose of the study is to assess the therapeutic education of patients with chronic respiratory failure who start to be treated with non invasive ventilation and during the first six months of ventilation.

DETAILED DESCRIPTION:
Therapeutic education about non invasive ventilation in patients with chronic respiratory failure and alveolar hypoventilation is assessed during the first six months of ventilation thanks to a questionnaire. Moreover, the impact of this therapeutic education on non invasive ventilation compliance, blood gas, dyspnea and nocturnal desaturation is assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic respiratory failure
* with alveolar hypoventilation required non invasive ventilation
* Adults and non-vulnerable subject
* Fluency in French

Exclusion Criteria:

* Age under eighteen years old
* Patient with guardianship
* No french-speaking
* Severe cognitive abnormalities
* No criteria to introduce non invasive ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Score efficacy of therapeutic education | 6 months
  calculation of the global mean score of the questionnaire dedicated to the knowledge about the ventilation device

SECONDARY OUTCOMES:
Compliance with the non invasive ventilation | 6 months
  number of hours of non invasive ventilation use per day
Dyspnea score | 6 months
  Dyspnea severity scoring between 0 and ten

CONTACTS AND LOCATIONS:
Locations (1):
- INSERM-UPC UMR_S 1158 Service de Pneumologie et Réanimation, R3S, Groupe Hospitalier Pitié-Salpêtrière, Paris, France